CLINICAL TRIAL: NCT05899582
Title: Extracranial-intracranial Bypass Surgery Versus Medical Treatment Alone for Symptomatic Chronic Middle Cerebral Artery Occlusion: the CMOSS-2 Trial
Brief Title: Extracranial-intracranial Bypass Surgery for Symptomatic Chronic Middle Cerebral Artery Occlusion: the CMOSS-2 Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMOSS-2
Record Dates: First submitted 2023-05-23; First posted 2023-06-12 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Symptomatic Chronic Middle Cerebral Artery Occlusion; Infarction, Middle Cerebral Artery
Keywords: middle cerebral artery occlusion; stroke; TIA
MeSH Terms: conditions — Infarction, Middle Cerebral Artery; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery (Experimental): The patients in the surgical group will be treated with direct extracranial to intracranial bypass surgery plus best medical treatment.
  Interventions: Procedure: Extracranial-Intracranial Bypass Surgery
- Medical treatment (Active Comparator): The patients will receive medical treatment alone according to the AHA/ASA Stroke and Transient Ischemic Attack (TIA) Stroke Prevention Guidelines (2021 edition).
  Interventions: Other: Medical treatment alone

INTERVENTIONS:
Procedure: Extracranial-Intracranial Bypass Surgery — Extracranial-intracranial bypass surgery plus medical treatment
  Arms: Surgery
Other: Medical treatment alone — Best medical treatment alone according to current clinical guidelines, including antiplatelet drugs (e.g. aspirin) and risk factor controls.
  Other Names: Best medical treatment
  Arms: Medical treatment

SUMMARY:
The CMOSS-2 trial is a government-funded, prospective, multicenter, randomized controlled trial. It will recruit symptomatic chronic occlusion of the middle cerebral artery in patients with severe hemodynamic insufficiency. Only high-volume center with a proven track record will be included. Patients will be randomized (1:1) to best medical treatment alone or medical treatment plus bypass surgery. Primary outcome is ischemic stroke in the territory of the target artery within 24 months after randomization.

DETAILED DESCRIPTION:
Middle cerebral artery occlusion is an important cause of ischemic stroke, and there are currently two treatment methods: medical treatment alone and extracranial-intracranial bypass surgery (EC-IC bypass surgery). Previous studies have shown that the optimal medical treatment has an annual stroke recurrence rate of up to 10%, and patients with concomitant hemodynamic disorders can also increase by 7.3 times.

The CMOSS study was the first trial in China to evaluate the safety and efficacy of EC-IC bypass surgery on patients with ICA or MCA occlusion combined with hemodynamic insufficiency evaluated with CT perfusion. The results showed that there was no significant difference in the risk of stroke or death between the bypass group and the medical group, but there was a significant difference in ipsilateral ischemic stroke between 30 days and 2 years after randomization, with only 2.0% in the surgery group and 10.3% in the medical group; In addition, subgroup analysis found that for patients with MCA occlusion or severe hemodynamic insufficiency, bypass surgery has a potential beneficial trend over medical treatment alone.

The CMOSS-2 trial is a government-funded, prospective, multicenter, randomized controlled trial. It will recruit symptomatic chronic occlusion of the middle cerebral artery in patients with severe hemodynamic insufficiency. Only high-volume center with a proven track record will be included. Patients will be randomized (1:1) to best medical treatment alone or medical treatment plus bypass surgery. Primary outcome is ischemic stroke in the territory of the target artery within 24 months after randomization. The CMOSS-2 trial will be conducted in 13 sites in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-65 years;
2. Confirmed as chronic occlusion of unilateral middle cerebral artery (MCA) by digital subtraction angiography (DSA) or computed tomography angiography (CTA). Other cerebral artery stenosis should be less than 50%.
3. CT perfusion demonstrates severe hemodynamic insufficiency in the territory of the qualifying MCA with MTT (symptomatic side) ≥ 6s or rCBF (symptomatic side/contralateral side) ≤ 0.8;
4. mRS score is 0-2 points;
5. A history of ischemic events (including<1/2 cerebral infarction in the middle cerebral artery supply area, or transient ischemic attack [TIA]) related to the qualifying artery within 12 months ;
6. The onset of acute stroke should be more than 1 month;
7. CT or MRI excludes large cerebral infarction (infarction>1/2 of the territory of the qualifying middle cerebral artery);
8. Patients or their guardians voluntarily participate of the study and sign the consent form.

Exclusion Criteria:

1. History of intracranial hemorrhage, subarachnoid hemorrhage, subdural hemorrhage, or extradural hemorrhage within 6 weeks;
2. Unstable angina pectoris or myocardial infarction, congestive heart failure within 6 months;
3. Women who are pregnant or lactating;
4. Coagulation dysfunction or hemorrhagic tendency (e.g. INR > 1.5 and/or platelet count < 100,000 mcL);
5. Other diseases with a life expectancy of less than 2 years
6. Previous treatment with EC-IC bypass surgery
7. Known allergy or contraindication to aspirin or clopidogrel or other antiplatelet drugs.
8. Known cardiac conditions that may lead to cardiogenic embolism: including prosthetic valves, infective endocarditis, left atrial or left ventricular thrombosis, atrial fibrillation, sick sinus node syndrome, atrial mucinous tumor or cardiomyopathy, ejection fraction <25%;
9. Allergy to iodine or x-ray contrast, blood creatinine > 3.0 mg/dl or other contraindications to arteriography
10. Uncontrolled diabetes mellitus with fasting blood sugar (FBS) >16.7 mmol/L
11. Uncontrolled hypertension with a sitting systolic blood pressure >180 mmHg or a sitting diastolic blood pressure >110 mmHg;
12. Persistent worsening of neurological symptoms within 72 hours;
13. Severe liver dysfunction, defined as serum alanine transaminase (ALT) and/or glutamic oxalacetic transaminase (AST) > 3 times the upper limit of normal range;
14. Active peptic ulcer disease;
15. Having received a clinical trial drug or device within 30 days prior to screening, or being enrolled in another clinical trial;
16. Other diseases or medical history that, in the judgment of the investigator, may affect the efficacy or safety evaluation of this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 420 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with ischemic stroke in territory of qualifying artery | 2 years after randomization
  Number of participants with ischemic stroke in territory of qualifying artery within 2 years after randomization

SECONDARY OUTCOMES:
Number of participants with any stroke or death | 30 days after randomization
  Number of participants with any stroke or death within 30 days after randomization
A composite of any stroke or death within 30 days, or ischemic stroke in territory of qualifying artery beyond 30 days to 2 years after randomization | within 2 years after randomization
  Number of participants with any stroke or death within 30 days, or ischemic stroke in territory of qualifying artery beyond 30 days to 2 years after randomization
Number of participants with any stroke | within 2 years after randomization
  Number of participants with any stroke within 2 years after randomization
Number of participants with disabling stroke (mRS>3) | within 2 years after randomization
  Number of participants with disabling stroke within 2 years after randomization
Number of participants with fatal stroke (death caused by a stroke) | within 2 years after randomization
  Number of participants with fatal stroke within 2 years after randomization
Number of participants with death | within 2 years after randomization
  Number of participants with death within 2 years after randomization
Number of participants with any stroke or death | within 2 years after randomization
  Number of participants with any stroke or death within 2 years after randomization
Functional outcomes of participants | 2 years after randomization
  Functional outcomes of participants such as modified Rankin scale (mRS) or the National Institutes of Health Stroke Scale (NIHSS) at 2 years after randomization
Anastomosis patency of participants in surgical group | 2 years after randomization
  Anastomosis patency of participants in surgical group at 2 years after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Jiao, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University., Beijing, China

IPD SHARING:
Plan to Share IPD: No